CLINICAL TRIAL: NCT05688930
Title: Effects of a Neuromuscular Training Program for the Prevention of Ankle Functional Instability in Male Soccer Players Aged 17-20: Randomized Clinical Trial With FIFA 11+
Brief Title: Effects of a Neuromuscular Training Ankle Preventive Program in Soccer Player
Acronym: PENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Manizales, Colombia (Other)
Collaborators: Universidad Católica del Maule (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 703-2020 T.D.
Record Dates: First submitted 2021-10-19; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Prevention and Control
Keywords: Ankle injuries; Physical therapy; Neuromuscular training; Functional ankle instability; Prevention; Unstable joint.
MeSH Terms: conditions — Ankle Injuries; Joint Instability | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: G1: Neuromuscular training program of prevention of functional ankle instability PEMNT; G2: FIFA 11+ Program Group (control).
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENMT (Experimental Group) (Experimental): The neuromuscular injury prevention intervention protocol contains field work activities that involve proprioceptive exercises, flexibility, and specific and general muscle strength of the MMII and trunk.
  Interventions: Other: PENMT (Experimental Group)
- FIFA 11+ (Control Group) (Active Comparator): Treatment or experimental condition. 1: FIFA 11+ Program
  Interventions: Other: FIFA 11+ (Control Group)

INTERVENTIONS:
Other: PENMT (Experimental Group) — The neuromuscular injury prevention intervention protocol contains field work activities that involve proprioceptive exercises, flexibility, and specific and general muscle strength of the MMII and trunk soccer players.
  Arms: PENMT (Experimental Group)
Other: FIFA 11+ (Control Group) — Treatment or experimental condition. 1: FIFA 11+ Program
  Arms: FIFA 11+ (Control Group)

SUMMARY:
Objetive:To determine the effects of a functional ankle instability prevention neuromuscular training (PENMT) program compared to the conventional FIFA 11+ program on the occurrence of ankle sprains, flexibility, balance and muscle activation in 17-year-old male youth soccer players to 20 years.

Subjects and Methods: An experimental investigation, controlled, randomized and single-blind clinical trial was carried out in 40 subjects randomized to start the control or experimental group (soccer Players). The trial compared the effects of a differential intervention with a protocol focused on an ankle neuromuscular training program vs the usual FIFA 11+ program, in order to strengthen functional ankle stability in youth soccer in male players. In each subject, 2 measurements were taken: Pre-intervention and Post-intervention. For each measurement, a hypothesis test was performed.

Results: The FIFA11+ is expressed as an injury risk factor when buying it with the PENMT after their participation.

Conclusion:The neuromuscular training program for the ankle or PENMT applied in the experimental group did not generate a negative effect with respect to the FIFA 11+ program, in addition to the time of departure in the post test, the PENMT program is expressed as a protection factor of player injuries when contrasted with the FIFA 11+ program, that is, it presents effectiveness against the risk factor of functional ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Be between the age range of 17 to 20 years old at the time of evaluation and intervention.
* Have a minimum of 2 years of semi-professional / professional sports practice.
* Be linked to the football club for at least 1 year.
* That they practice soccer at least 5 times a week.
* That they are playing at least one competitive tournament.
* That they have an active or current health promotion entity - EPS and / or occupational risk insurer-ARL.
* Players who during the entire period of 2019-2020 have presented at least one episode of lateral ankle sprain (during the last 4 months) (in the time range of 3 to 12 months prior to the first evaluation) who have required immobilization and / or weight loss for at least 3 days; present pain, subjective perception questionnaires of ankle instability).
* Soccer players with or without sprained ankle injuries will be taken, but not in the last 3 months. However, the time elapsed since the last episode will be recorded.

Exclusion Criteria:

* Belonging to another sports club and / or regularly practicing more than one sport with muscular demand of the lower tract (lower limbs).
* Who present acute injuries such as: vestibular alterations, history of ankle fracture, acute knee and / or ankle injury during the last 3 months, history of previous surgical interventions in lower limbs or underlying systemic disease at the time of the initial evaluation (pretest).
* Who are undergoing treatment for any neuromuscular or other related pathology, in the acute phase and / or who have received a neuromuscular training program in the last 4 months, different from the one that will be applied in this study.
* That in the last 4 months they have been in treatment for any neuromuscular pathology or other related to the acute phase and / or receive a neuromuscular training program different from the one that will be applied in this study.

Ages: 17 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Preventive program (Type of) | 12 weeks
  Neuromuscular and functional training protocol

SECONDARY OUTCOMES:
Ankle instability perception | Two measurements: first week and twelfth week
  Two measures were performed for each patient; Cumberland Ankle Instability Questionnaire (CAIT): 30 points no instability; less than 27 points presence of ankle instability. (applied pre and post intervention moments)
Measurement flexibility (centimeters) | Two measurements: first week and twelfth week
  Two measures were performed for each patient; of the ankle joint (Lunge test) and chain of the lower limb (sit and reach: (BSSR); measurement in centimeters (cm), report of negative values or less than 0 cm, presence of retraction was lost. Both before and after the test.(applied pre and post intervention moments)
Limits of stability - balance (millimeters) | Two measurements: first week and twelfth week
  Two measures were performed for each patient;Dynamic and static balance with eyes open and closed, in a movement analysis laboratory, measured in millimeters -mm. (Applied moments pre and post intervention)
Measured with conduction velocity in seconds under maximal voluntary contraction (MVC) | Two measurements: first week and twelfth week
  Two measures were performed for each patient; surface electromyography, musculature - at 25 percentage, 50 percentage and 75 percentage of muscle activation. (moments before and after the intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Lina Ma Montealegre, Msc, Principal Investigator — U.AUTÓNOMA
Locations (1):
- Autonoma's University, Manizales, Caldas Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brito J, Malina RM, Seabra A, Massada JL, Soares JM, Krustrup P, Rebelo A. Injuries in Portuguese youth soccer players during training and match play. J Athl Train. 2012 Mar-Apr;47(2):191-7. doi: 10.4085/1062-6050-47.2.191. PMID 22488285
- [Background] Imai A, Imai T, Iizuka S, Kaneoka K. A Trunk Stabilization Exercise Warm-up May Reduce Ankle Injuries in Junior Soccer Players. Int J Sports Med. 2018 Apr;39(4):270-274. doi: 10.1055/s-0044-100923. Epub 2018 Feb 15. PMID 29448292
- [Background] Halasi T, Kynsburg A, Tallay A, Berkes I. Changes in joint position sense after surgically treated chronic lateral ankle instability. Br J Sports Med. 2005 Nov;39(11):818-24. doi: 10.1136/bjsm.2004.016527. PMID 16244190